CLINICAL TRIAL: NCT06342739
Title: Verbal Synchrony, Satisfaction and Decision-making in Face-to-face Consultations
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1595
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Benign thyroid nodules group: Participants with benign thyroid nodules involved in a consultation with endocrinologist and/or surgeon and/or radiologist, in order to discuss treatment options related to benign thyroid nodules

SUMMARY:
Eligible participants will be: benign thyroid nodules patients, to be involved in a consultation with their endocrinologist and/or surgeon and/or radiologist, in order to discuss treatment options related to benign thyroid nodules.

DETAILED DESCRIPTION:
Eligible participants will be: benign thyroid nodules patients, to be involved in a consultation with their endocrinologist and/or surgeon and/or radiologist, in order to discuss treatment options related to benign thyroid nodules. Endocrinologist and/or surgeon and/or radiologist involved in the consultation will be recruited as well.

Before the scheduled consultation with endocrinologist, surgeon or radiologist, benign thyroid nodules patients will be screened for eligibility by a researcher and a physician from the Interventional Radiology Unit.

If patients meet all the inclusion criteria, they will be contacted by the researcher and proposed to participate. The day of the consultations, researcher will meet participants face to face, they will answer any questions should arise and will ask them to sign the informed consent form.

Benign thyroid nodules patients have a specific clinical pathway, in which they may have consultations with endocrinologists, and/or with surgeon, and/or with radiologists. Patients will be recruited before their first consultation and then, if they are scheduled to have other consultations with other professionals, will be recruited as well for the following consultations.

ELIGIBILITY:
Inclusion Criteria:

Specifically, to be eligible for the inclusion in this study, each patient has to fulfill all these criteria:

* diagnosis of benign thyroid nodule;
* scheduled consultation with endocrinologist and/or surgeon and/or radiologist to discuss treatment options related to benign thyroid nodule;
* ≥18 years old at the time of recruitment;
* proper understanding of Italian language;
* fluent Italian speaker;
* able to comply to requested procedures to obtain audio-video recording.

Each professional has to fulfill these criteria:

* proper understanding of Italian language;
* fluent Italian speaker;
* able to comply to requested procedures to obtain audio-video recording.

Exclusion Criteria:

• Patients with diagnosed mental or neurological disorder that could impair the participation will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of benign thyroid nodule with a scheduled consultation with endocrinologist and/or surgeon and/or radiologist to discuss treatment options related to benign thyroid nodule at European Institute of Oncology
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of predictive power of verbal synchrony established between patient and physician during the consultation on patients' satisfaction | 1 month
  The primary endpoint of our research is to test the predictive power of verbal synchrony established between patient and physician during the consultation on patients' satisfaction with tha analysis of audio and video recording file.
  Variables analyzed from audio recording will be use of words, verbal synchrony, empathic communication; variables analyzed from video recording will be facial emotion expression and facial emotion expression synchrony

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy